CLINICAL TRIAL: NCT06853054
Title: A New Approach to Vascular Reconstruction Using Graphical 3D Printing and Flow Modelling to Create Personalized Precision Engineered Surgery
Brief Title: Seeking for Perfected Aortic Arch Reconstruction Using a Graphically Designed Patient-specific Surgical Patch
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Shi-Joon Yoo, Staff Cardiac Radiologist, Division of Cardiac Imaging, Department of Diagnostic Imaging, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1000081239
Record Dates: First submitted 2024-11-07; First posted 2025-02-28 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Hypoplastic Left Heart Syndrome (HLHS); Aortic Arch Hypoplasia
Keywords: Congenital heart surgery; Aortic arch reconstruction; Surgical patch; Computer-aided design; 3D modeling and printing
MeSH Terms: conditions — Hypoplastic Left Heart Syndrome

STUDY DESIGN:
Intervention Model Description: Feasibility study to obtain preliminary data on the surgical outcomes (clinical hemodynamics, procedural times, reconstructed aortic arch configuration, geometry and size) of patients using traditional versus personalized patches.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Personalized Patch Template (Experimental): Using each participant's pre-operative imaging, the most ideal aortic arch configuration will be identified. This will be followed by simulation of mechanical effects on the adjacent structures by overlapping the designed aortic arch model on the participant's original images. Computer-aided design of the personalized patch template will then be completed and followed by 3D printing of the sterilizable, personalized patch template.
  Interventions: Procedure: Personalized patch template

INTERVENTIONS:
Procedure: Personalized patch template — The personalized, sterilizable patch template will be used as the surgeon's guide in fashioning the precise size and shape of the surgical patch.

SUMMARY:
Vascular Reconstruction is one of the most challenging areas of surgery, the surgeon has to create a completely watertight reconstruction without any narrowing or deformity that will restore normal flow characteristics, even at high pressures. Nowhere is this more challenging than in neonatal heart surgery where babies born with aortic arch narrowing or underdevelopment are one of the commonest life-threatening cardiovascular conditions.

Reconstruction not only has to recreate normal anatomy but also allow for subsequent growth and development.

Until now, surgical reconstruction depended on the surgeon's subjective assessment of the anatomy and a best estimate of patch shaping and design. New engineering techniques have enabled us to create 3D printed models of real hearts and then recreate the actual surgery on these models using a variety of engineered patches and different surgical techniques. These reconstructed models can now be placed in flow-testing rigs and undergo 4-dimensional flow imaging to provide high-fidelity velocity and shear force analysis that allow for precision design of the ideal geometry to give optimal flow.

This project will combine the skills of the largest team of neonatal heart surgeons in Canada, working with cardiac imaging experts, physicists and biomechanical engineers who are recognized as the world leaders in 3D printing technologies for congenital heart disease. Using a series of rigorous repeated tests and different designs we will define the ideal techniques and patch shapes and then translate this to real cases where a precision-shaped personalized patch can be created for each individual. Following up these babies as they grow with precision 3D scanning will show how these vessels are growing. Our mathematics-driven approach will make the surgery easier, shorter and more efficient. It will also provide more consistent surgical results among surgeons.

DETAILED DESCRIPTION:
Aortic arch reconstruction complications can be prevented or minimalized by personalizing the surgical technique and patch through mathematical computer modeling and 3D printing.

This is a feasibility study on the use of graphical 3D printing and flow modelling in the creation of personalized patch templates for the Norwood procedure and aortic arch reconstruction.

Patients undergoing the Norwood procedure as part of standard of care will be approached for consent. Patients who consent to the study will undergo a pre-operative contrast CT scan to design simulation models and to identify the most ideal aortic arch configuration. 3D printing of the sterilizable template will be done after computer-aided design of bespoke surgical patches and will be based on pre-operative imaging and simulation. The sterilizable patch template will be used by the surgeon as a guide to fashioning the precise size and shape of the patch.

A research CT scan will be done post-operatively, prior to patient discharge. The post-op CT scan will be used to create a 3D printed model of the reconstructed aortic arch, This 3D printed model will then undergo 4D MRI scanning as part of the analysis.

Patients will be monitored and followed closely post-surgery. They will be assessed by routine post-operative tests including standard of care imaging at 4-6 months after surgery.

Clinical outcome assessment at 6-12 months after surgery will be measured.

This data will be compared to surgical outcomes of a historical cohort of patients who had traditional patches.

ELIGIBILITY:
Inclusion Criteria:

* Newborns, 0-2 months of age
* Requiring a Norwood procedure and aortic arch reconstruction
* Consent provided

Exclusion Criteria:

* Consent not provided
* Contraindications to contrast CT scans (allergy to contrast, kidney disease)
* Any condition or diagnosis, that could in the opinion of the Principal Investigator or delegate interfere with the participant's ability to comply with the study, might confound the interpretation of the study results, or put the participant at risk

Ages: 0 Months to 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Survival Rate (%): patient status (Alive/Dead) | In hospital, at 30 days and at 1 year follow-up
  Survival will be recorded based on patient status at the time of discharge (in-hospital), 30 days post-surgery, and at 1-year follow-up. The unit of measure will be the percentage of patients who remain alive at each of these time points.
Hemodynamic Stability: Inotrope Requirement (daily score) | Post-op Day 1: Initial assessment within 24 hours of surgery, Post-op Days 2-7: Daily assessments during the first week post-surgery, 1 month, 6 months, 1 year follow up: Evaluation of ongoing hemodynamic stability
  A scale measuring the need for inotropic support, based on the number and type of inotropic medications required. Inotropic support will be quantified on a daily score (ranging from 0 to a maximum score depending on inotrope usage).
Hemodynamic Stability: Blood pressure | Post-op Day 1: Initial assessment within 24 hours of surgery, Post-op Days 2-7: Daily assessments during the first week post-surgery, 1 month, 6 months, 1 year follow up: Evaluation of ongoing hemodynamic stability
  Measured in mmHg using a standard non-invasive sphygmomanometer or an arterial catheter for continuous measurement in the ICU.
Hemodynamic Stability: Heart Rate | Post-op Day 1: Initial assessment within 24 hours of surgery, Post-op Days 2-7: Daily assessments during the first week post-surgery, 1 month, 6 months, 1 year follow up: Evaluation of ongoing hemodynamic stability
  Measured in beats per minute (bpm) using ECG or pulse oximeter.
Hemodynamic Stability: Oxygen Saturations (SpO2) | Post-op Day 1: Initial assessment within 24 hours of surgery, Post-op Days 2-7: Daily assessments during the first week post-surgery, 1 month, 6 months, 1 year follow up: Evaluation of ongoing hemodynamic stability
  Measured as a percentage (%) using a pulse oximeter.

SECONDARY OUTCOMES:
Need for Re-intervention or Additional Surgeries (%) | During hospitalization, at 1 Month, 6 Months, and 1 Year Follow-up
  Patient status (Need for re-exploration, reoperation, or catheter-based interventions) measured by the percentage (%) of patients requiring additional surgical or catheter-based interventions.
Incidence of Post-operative Complications (%) | Post-op Days 1-3, Post-op days 4-7, Post Discharge (1 month, 6 months, 1 year)
  Percentage (%) of patients with complications (e.g., renal dysfunction, infection, bleeding, metabolic distress)
Growth Parameters at Follow-up: Weight | At hospital discharge, at 1 Month, 6 Months, and 1 Year follow-up
  Measurement of weight in kg
Growth Parameters at Follow-up: Height | At hospital discharge, at 1 Month, 6 Months, and 1 Year follow-up
  Measurement of height (cm)
Growth Parameters at Follow-up: Oxygen saturation in % | At hospital discharge, at 1 Month, 6 Months, and 1 Year follow-up
  Measurement of oxygen saturation SpO2 (%)
Aortic Arch Dimensions (mm) | At pre-op, post-op day 1, and at follow-up: a 1 month, 6 months and 1 year post surgery
  Aortic arch dimensions in mm (measured in different sections of the arch: ascending aorta, proximal, distal, isthmus).
Flow velocity | At pre-op, post-op day 1, and at follow-up: a 1 month, 6 months and 1 year post surgery
  Flow velocity in cm/s (measured using Doppler ultrasound or MRI 4D flow study).
Cardiac Function (Ventricular Function and Valve Regurgitation) and Heart Structure (Atrial Septum Integrity) | At pre-op, post-op day 1, and at follow-up: a 1 month, 6 months and 1 year post surgery
  Qualitative assessment of ventricular function, the atrial septum, tricuspid regurgitation and neo-aortic regurgitation through echocardiography
Long-term Reintervention or Complications | At 1 month, 6 months, and 1 year follow-up
  Percentage (%) of patients requiring reintervention or experiencing complications
Incidence of Structural Issues (Pulmonary or Bronchial Compression) (%) | At post-op Day 1 and at 1 month, 6 months and 1 year follow-up
  Percentage (%) of patients with left pulmonary artery compression, left main bronchus compression, or aortic arch tortuosity as measured by CT or MRI scans.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No